CLINICAL TRIAL: NCT03167658
Title: The Impact of Employee Wellness Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Robert Wood Johnson Foundation (Other); National Institute on Aging (NIA) (NIH); Abdul Latif Jameel Poverty Action Lab (Other); University of Chicago (Other)
Responsible Party: Principal Investigator, Zirui Song, Assistant Professor of Health Care Policy and Medicine, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Wellness 14-3141; R01AG050329 (NIH); P30AG012810 (NIH); 72611 (Other Grant/Funding Number: Robert Wood Johnson Foundation); AEARCTR-0000586 (Registry Identifier: American Economic Association Trial Registry)
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Health Behavior; Disease, Chronic
Keywords: Wellness; Prevention
MeSH Terms: conditions — Health Behavior; Chronic Disease

STUDY DESIGN:
Intervention Model Description: Each worksite (and all employees at that site) randomly assigned to Treatment or Control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment (Experimental): Employees at treatment worksites will be given access to workplace wellness programming. Participation by employees will be voluntary, but all employees at treatment sites will be considered as part of the treatment group. Employees will also be invited to complete on-site biometric assessments and questionnaires. Data from secondary data sources (including employment records and health insurance claims) will be collected for employees at all BJ's worksites.
  Interventions: Behavioral: Workplace wellness program
- Primary Control (No Intervention): Employees at primary control worksites will be invited to complete on-site biometric assessments and questionnaires, but will not have access to the workplace wellness programming. Data from secondary data sources (including employment records and health insurance claims) will be collected for employees at all BJ's worksites.
- Secondary Control (No Intervention): Employees at secondary control worksites will not participate in in-person screenings or questionnaires, and will not have access to workplace wellness programming. Data from secondary data sources (including employment records and health insurance claims) will be collected for employees at all BJ's worksites.

INTERVENTIONS:
Behavioral: Workplace wellness program — Multi-prong workplace wellness program, with components such as nutrition counseling, fitness challenges, and stress management workshops, including supports and incentives.
  Arms: Treatment

SUMMARY:
There is great public and private interest in the use of workplace wellness programs to reduce health care spending, improve health outcomes, and enhance productivity for employees. However, there is little rigorous evidence on the effects of wellness programs. This study partners with a large multi-state U.S. employer (BJ's Wholesale Club) and an experienced wellness vendor (Wellness Workdays) to evaluate a multi-prong workplace wellness program, including components such as nutrition counseling, fitness challenges, and stress management workshops. The wellness program will be delivered by a team of experts including Registered Dieticians, and will include financial rewards for participation. The program will be available to employees in initially 20 of BJ's 200 worksites, and later expanded to 25 worksites. These worksites have been randomly selected, allowing a randomized controlled trial evaluation of the effects of the wellness program. Data will be collected on a wide array of outcomes from multiple sources, including on-site biometric screenings and surveys, employment records, and health insurance claims for employees at both treatment and control worksites.

ELIGIBILITY:
Inclusion Criteria:

* Employed in one of BJ's clubs during the period of the intervention

Exclusion Criteria:

* Not employed in one of BJ's clubs during the period of the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48664 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Physical activity | Primary data collected at 18 months and 30 months after initiation of intervention
  Regular exercise, number of hours sitting per day, and actively managing weight, as indicated in responses to survey questions
Obesity | Primary data collected at 18 months and 30 months after initiation of intervention
  Body Mass Index>=30, calculated from measured height and weight
Absenteeism | Administrative records from 3 years spanning intervention
  Number of sick or personal days as a share of total days employed, from employment records
Health care spending | Administrative records from 3 years spanning intervention
  Dollars spent on health care for employees covered by employer-sponsored insurance, from claims records

OTHER OUTCOMES:
Blood pressure | Primary data collected at 18 months and 30 months after initiation of intervention
  Systolic blood pressure, measured
Depression | Primary data collected at 18 months and 30 months after initiation of intervention
  Unmanaged depression, as indicated in responses to survey questions
Tenure | Administrative records from 3 years spanning intervention
  Duration of employment in days, from employment records
Job performance | Administrative records from 3 years spanning intervention
  Numerical performance rating from annual review, from employment records
Health care spending (i.e. dollars spent) | Administrative records from 3 years spanning intervention
  Dollars spent on health care and prescription drugs for employees covered by employer-sponsored insurance, decomposed into spending on inpatient, outpatient, emergency department, and prescription drugs, from claims records
Health care utilization (i.e. number of doctor visits, hospitalizations, or medications) | Administrative records from 3 years spanning intervention
  Health care encounters and prescription drugs for employees covered by employer-sponsored insurance, decomposed into inpatient, outpatient, emergency department, and prescription drugs, from claims records
Nutrition management | Primary data collected at 18 months and 30 months after initiation of intervention
  Affirmative engagement in active efforts to improve nutrition, as indicated in responses to survey questions
Stress management | Primary data collected at 18 months and 30 months after initiation of intervention
  Unmanaged stress and stress at work, as indicated in responses to survey questions
Screenings and exams | Primary data collected at 18 months and 30 months after initiation of intervention
  Percent of recommended tests received, as indicated in responses to survey questions
Tobacco use | Primary data collected at 18 months and 30 months after initiation of intervention
  Smoking, as indicated in responses to survey questions
Health and wellbeing | Primary data collected at 18 months and 30 months after initiation of intervention
  Short form 8 (SF-8) physical and mental summary scores, as indicated in responses to survey questions. Each question of the SF-8 uses a 5- or 6-point Likert scale. Its standardized scoring system combines responses into a score that can be interpreted as a continuous variable (analogous to a 0-100 scale), with higher scores denoting better self-reported health.
Blood glucose | Primary data collected at 18 months and 30 months after initiation of intervention
  Blood glucose, measured
Cholesterol | Primary data collected at 18 months and 30 months after initiation of intervention
  Total cholesterol and high-density lipoprotein (HDL), measured

CONTACTS AND LOCATIONS:
Overall Officials: Zirui Song, MD, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Song Z, Baicker K. Effect of a Workplace Wellness Program on Employee Health and Economic Outcomes: A Randomized Clinical Trial. JAMA. 2019 Apr 16;321(15):1491-1501. doi: 10.1001/jama.2019.3307. PMID 30990549

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/58/NCT03167658/Prot_SAP_001.pdf